CLINICAL TRIAL: NCT06093022
Title: Surgical or Medical Treatment of Breast Cancer Metastasis: A Multicentre Observational Study
Acronym: SurMed-BCLM
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5795
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Liver Metastases
Keywords: breast cancer; liver metastasis; liver surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BCLM-surg: BCLM underwent liver resection
- BCLM-med: BCLM underwent medical treatment alone

SUMMARY:
The liver represents the third most common site of breast cancer (BC) metastases behind the lymphatics and bone. The primary treatment for BCLM remains chemo-therapy and, more recently, targeted immunotherapy. The role of liver resection in BCLM remains controversial. The primary aim of the study is to compare the efficacy of liver resection vs. medical therapy alone in Breast Cancer Liver Metastasis (BCLM) patients.

DETAILED DESCRIPTION:
In this multicenter observational ambispective study, will be enrolled all patients with BCLM underwent liver resection or medical treatment alone afferent to the Fondazione Policlinico Gemelli IRCSS of Rome (Italy), and other 8 International centers

The study foresees two distinct phases:

* I phase (only retrospective phase): it will cover all patients underwent to either medical treatment or surgery for which all data are available, with a follow up of 5 years at March 31, 2023. All patients data will be recovered from January 1994 till March 31, 2018. At the end of "phase I", is provided an "ad interim" analysis.
* II phase (ambispective): All patients retrieved from the archives between April 1, 2018 and the April 30, 2023 will be included, as well as all prospectively enrolled patients till December 31 2023, so that the last patient enrolled will end the 5-years follow-up phase within December 31, 2028.

The primary endpoint is to analyze the efficacy of liver surgery as compared to medical therapy alone in terms of 5-years overall survival in patients with breast cancer who underwent to liver resection or medical therapy alone.

The secondary endpoints are: recurrence rate; post-operative mortality (in patients who underwent to surgical treatment), post-operative complication (in patients who underwent to surgical treatment). And also: to assess potential predictive factors of 5-years overall survival in patients with breast cancer who underwent to either liver resection or medical therapy alone, to assess recurrence free survival (RFS) of liver surgery as compared to medical therapy alone in terms of 5-years overall survival in patients with breast cancer who underwent to liver resection or medical therapy alone and to assess potential predictive factors of 5-years RFS in patients with breast cancer who underwent to either liver resection or medical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* BCLM
* BCLM and extra-hepatic disease
* Any treatment
* Ability to understand and sign the informed consent

Exclusion Criteria:

* Inability to provide the informed consent
* Patient who underwent Best Supportive Care or Palliation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with BCLM underwent liver resection or medical treatment alone.
Sampling Method: Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
5-years overall survival | 2018-2023
  The efficacy of liver surgery as compared to medical therapy alone in terms of 5-years overall survival in patients with breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diamond JR, Finlayson CA, Borges VF. Hepatic complications of breast cancer. Lancet Oncol. 2009 Jun;10(6):615-21. doi: 10.1016/S1470-2045(09)70029-4. PMID 19482250
- [Background] Arciero CA, Guo Y, Jiang R, Behera M, O'Regan R, Peng L, Li X. ER+/HER2+ Breast Cancer Has Different Metastatic Patterns and Better Survival Than ER-/HER2+ Breast Cancer. Clin Breast Cancer. 2019 Aug;19(4):236-245. doi: 10.1016/j.clbc.2019.02.001. Epub 2019 Feb 14. PMID 30846407
- [Background] Ma R, Feng Y, Lin S, Chen J, Lin H, Liang X, Zheng H, Cai X. Mechanisms involved in breast cancer liver metastasis. J Transl Med. 2015 Feb 15;13:64. doi: 10.1186/s12967-015-0425-0. PMID 25885919
- [Background] DeSantis CE, Ma J, Gaudet MM, Newman LA, Miller KD, Goding Sauer A, Jemal A, Siegel RL. Breast cancer statistics, 2019. CA Cancer J Clin. 2019 Nov;69(6):438-451. doi: 10.3322/caac.21583. Epub 2019 Oct 2. PMID 31577379
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Howlader M, Heaton N, Rela M. Resection of liver metastases from breast cancer: towards a management guideline. Int J Surg. 2011;9(4):285-91. doi: 10.1016/j.ijsu.2011.01.009. Epub 2011 Jan 31. PMID 21281746
- [Background] Golse N, Adam R. Liver Metastases From Breast Cancer: What Role for Surgery? Indications and Results. Clin Breast Cancer. 2017 Jul;17(4):256-265. doi: 10.1016/j.clbc.2016.12.012. Epub 2017 Jan 9. PMID 28196771
- [Background] Rashid NS, Grible JM, Clevenger CV, Harrell JC. Breast cancer liver metastasis: current and future treatment approaches. Clin Exp Metastasis. 2021 Jun;38(3):263-277. doi: 10.1007/s10585-021-10080-4. Epub 2021 Mar 6. PMID 33675501
- [Background] Sadot E, Lee SY, Sofocleous CT, Solomon SB, Gonen M, Kingham TP, Allen PJ, DeMatteo RP, Jarnagin WR, Hudis CA, D'Angelica MI. Hepatic Resection or Ablation for Isolated Breast Cancer Liver Metastasis: A Case-control Study With Comparison to Medically Treated Patients. Ann Surg. 2016 Jul;264(1):147-154. doi: 10.1097/SLA.0000000000001371. PMID 26445472
- [Background] Ruiz A, van Hillegersberg R, Siesling S, Castro-Benitez C, Sebagh M, Wicherts DA, de Ligt KM, Goense L, Giacchetti S, Castaing D, Morere J, Adam R. Surgical resection versus systemic therapy for breast cancer liver metastases: Results of a European case matched comparison. Eur J Cancer. 2018 May;95:1-10. doi: 10.1016/j.ejca.2018.02.024. Epub 2018 Mar 23. PMID 29579478
- [Background] Mariani P, Servois V, De Rycke Y, Bennett SP, Feron JG, Almubarak MM, Reyal F, Baranger B, Pierga JY, Salmon RJ. Liver metastases from breast cancer: Surgical resection or not? A case-matched control study in highly selected patients. Eur J Surg Oncol. 2013 Dec;39(12):1377-83. doi: 10.1016/j.ejso.2013.09.021. Epub 2013 Oct 6. PMID 24126165
- [Background] Lakatos E. Designing complex group sequential survival trials. Stat Med. 2002 Jul 30;21(14):1969-89. doi: 10.1002/sim.1193. PMID 12111882
- [Background] Schemper M, Wakounig S, Heinze G. The estimation of average hazard ratios by weighted Cox regression. Stat Med. 2009 Aug 30;28(19):2473-89. doi: 10.1002/sim.3623. PMID 19472308
- [Background] van Smeden M, Moons KG, de Groot JA, Collins GS, Altman DG, Eijkemans MJ, Reitsma JB. Sample size for binary logistic prediction models: Beyond events per variable criteria. Stat Methods Med Res. 2019 Aug;28(8):2455-2474. doi: 10.1177/0962280218784726. Epub 2018 Jul 3. PMID 29966490
- [Background] Moons KG, Altman DG, Reitsma JB, Ioannidis JP, Macaskill P, Steyerberg EW, Vickers AJ, Ransohoff DF, Collins GS. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): explanation and elaboration. Ann Intern Med. 2015 Jan 6;162(1):W1-73. doi: 10.7326/M14-0698. PMID 25560730

DOCUMENTS (2):
  • Study Protocol (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT06093022/Prot_000.pdf
  • Informed Consent Form (2023-04-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT06093022/ICF_001.pdf